CLINICAL TRIAL: NCT05492279
Title: Effect of Sheep Ghee on Lipid Profile and High-sensitivity C-reactive Protein: A Randomized Clinical Trial
Brief Title: Is Sheep Ghee Cardioprotective?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Kojuri, professor, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 98-01-01-22054
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Cholesterol; Metabolic Disorder; Inflammation
Keywords: Atherosclerosis; cardiovascular disease; high-sensitivity C-reactive protein; inflammation; sheep ghee
MeSH Terms: conditions — Metabolic Diseases; Inflammation; Atherosclerosis; Cardiovascular Diseases | interventions — Sunflower Oil

STUDY DESIGN:
Intervention Model Description: clinical trial randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: random allocation, open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): 10 gr Sheep ghee
  Interventions: Dietary Supplement: sheep ghee
- control group (Active Comparator): 10 gr sunflower oil
  Interventions: Dietary Supplement: sunflower oil

INTERVENTIONS:
Dietary Supplement: sheep ghee — natural sheep ghee, given to patient in a commercial box and intervention group 10 gr per day from sheep ghee
  Arms: intervention
Dietary Supplement: sunflower oil — natural sunflower oil, given to patients in a commercial box and patient use 10 gr of it
  Arms: control group

SUMMARY:
Normal volunteers were randomly received Sheep ghee or sunflower oil, and before and after the study lipid profile and HS-CRP were measured.

DETAILED DESCRIPTION:
During outpatient clinic visits, potentially eligible individuals were screened for enrollment according to the inclusion and exclusion criteria.

Patients were randomly allocated into the treatment and control groups via the blocked randomization method.

The control group received a normal diet for eight weeks with 10 g of sunflower oil. In the treatment group, sunflower oil was replaced with 10 g of sheep ghee.

50 patients in each group were enrollment. Patients' information, including demographic data and the serum levels of fasting blood sugar (FBS), LDL, HDL, triglyceride (TG), and hs-CRP, were recorded in datasheets twice: once before treatment with sheep ghee and once eight weeks later.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults, seeking outpatient visit at professor kojuri cardiology clinic

Exclusion Criteria:

* any history of ischemic heart disease (IHD),
* coronary artery bypass grafting (CABG)
* percutaneous intervention (PCI)
* stroke
* peripheral vascular diseases
* use of anti-hyperlipidemic agents
* unwillingness to participate.
* Need of tight hyperlipidemia control.

Ages: 20 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol | 2 months
  serum LDL level in mg/dl
total cholesterol | 2 months
  serum total cholesterol in mg/dl
HDL cholesterol | 2 months
  Serum HDL in mg/dl
HS-CRP | 2 months
  HS-CRP level in picogram/dl

SECONDARY OUTCOMES:
adverse effect | 2 months
  gastrointestinal, skin, allergy

CONTACTS AND LOCATIONS:
Locations (1):
- Javad Kojuri, Shiraz, Fars, Iran